CLINICAL TRIAL: NCT00404105
Title: A Prospective, Randomised Trial of Photo-Refractive Keratectomy (PRK) and Laser-in-Situ-Keratomileusis (LASIK) for Correction of Myopia
Brief Title: A Comparison of PRK and LASIK for Correction of Myopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUH-Ophthalmology-1999-01
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2006-11-27 (Estimated); Status verified 2006-11

CONDITIONS: Myopia
Keywords: Excimer laser
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

INTERVENTIONS:
Procedure: PRK
Procedure: LASIK

SUMMARY:
The study compares the precision and accuracy of two laser refractive techniques, PRK and LASIK, for correction of nearsightedness between -6 and -8 diopters.

ELIGIBILITY:
Inclusion Criteria:

* spherical equivalent subjective refraction between -6.00 and -8.00 diopters
* age between 18 and 49 years
* desire for having laser refractive surgery

Exclusion Criteria:

* present or past eye disease excluding myopia
* pregnant or lactating woman

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2000-06; Study Completion 2004-05

PRIMARY OUTCOMES:
Uncorrected visual acuity
Best corrected visual acuity
Best spectacle correction

SECONDARY OUTCOMES:
IOP
Corneal thickness
Corneal wavefront aberrations

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Hjortdal, MD, PhD, Principal Investigator — Department of Ophthalmology, Aarhus Sygehus, University of Aarhus
Locations (1):
- Department of Ophthalmology, Aarhus Sygehus NBG, Aarhus C, Denmark

REFERENCES:
- [Derived] Ivarsen A, Hjortdal J. Seven-year changes in corneal power and aberrations after PRK or LASIK. Invest Ophthalmol Vis Sci. 2012 Sep 6;53(10):6011-6. doi: 10.1167/iovs.12-10208. PMID 22879417